CLINICAL TRIAL: NCT00268567
Title: Phase 3 Study of Leflunomide Combined With Prednisone Treatment of Proliferative Lupus Nephritis as Induction Therapy
Brief Title: Induction Treatment of Proliferative Lupus Nephritis With Leflunomide Combined With Prednisone
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Peking University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLLNT-2002HL0133
Record Dates: First submitted 2005-12-21; First posted 2005-12-22 (Estimated); Last update posted 2005-12-22 (Estimated); Status verified 2004-10

CONDITIONS: Nephritis, Lupus
MeSH Terms: conditions — Lupus Nephritis | interventions — Prednisone

INTERVENTIONS:
Drug: leflunomide combined with prednisone

SUMMARY:
lupus nephritis accounts for the most morbidity and mortality in patients with SLE. Glucocorticoids combined with cyclophosphamide (CYC) are effective for the treatment of patients with proliferative lupus nephritis and have been the immunosuppressive regimen of choice for many years. However, some patients do not respond well to the regimen, and adverse effects of cyclophosphamide limit its use in certain patients. Leflunomide is a novel immunosuppressive agent currently used in the treatment of rheumatoid arthritis.There were a few pilot observational studies and reports suggesting leflunomide was also safe, well-tolerated and may be effective in SLE patients without important organ involvement. It has not been shown if leflunomide can be used in the treatment of patients with lupus nephritis. We therefore undertook a multi-center, controlled study to investigate the efficacy and safety profile of leflunomide compared with cyclophosphamide in the treatment of patients with biopsy proven proliferative lupus nephritis.

ELIGIBILITY:
Inclusion Criteria:

* All patients were diagnosed as SLE according to the updated criteria of American College of Rheumatology in 1997, had a systemic lupus erythematosus disease activity index (SLEDAI)equal or greater than 8; had evident renal diseases and biopsy-documented diffuse proliferative or focal proliferative lupus nephritis, with or without coincident membranous nephropathy, and pathological activity index (AI)equal or greater than 4

Exclusion Criteria:

* Patients who had received cyclophosphamide within the previous 3 months, cerebral lupus, severe infection, liver disease, pregnancy, and anticipated poor compliance with the protocol.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-10

PRIMARY OUTCOMES:
complete remission of renal disease at 6 months

SECONDARY OUTCOMES:
partial remission at 6 months and adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Wang, M.D., Principal Investigator — Institute of Nephrology, Peking University
Locations (8):
- China (8):
  - Renal Division, Peking University First Hospital, Beijing
  - Department of Nephrology, Kidney Center and key Lab of PLA, Chinese General Hospital of PLA, Beijing
  - Division of Nephrology, Nanfang Hospital, Southern Medical University, Guangzhou
  - Renal Division, the First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Department of Rheumatology, the Second Affiliated Hospital, Harbin Medical University, Harbin
  - Department of Nephrology, Shanghai Changzheng Hospital, Shanghai
  - Renal Division, Huashan Hospital, Fudan University, Shanghai
  - Renal Division, Renji Hospital, Shanghai Jiaotong University, Shanghai